CLINICAL TRIAL: NCT05550415
Title: Vimentin Expression-based Therapeutic Response in Triple Negative Breast Cancer Receiving Combination of Simvastatin and NAC: a Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Role of Simvastatin in the Epithelial-Mesenchymal Transition Process of Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. dr. Erwin Danil Yulian, Sp.B (K) Onk, Head of Research Program, Division of Surgical Oncology, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IndonesiaU2022
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Triple Negative Breast Cancer; Chemotherapy Effect; Simvastatin Adverse Reaction
Keywords: Vimentin; Simvastatin; Epithelial-Mesenchymal Transition; Neoadjuvant Chemotherapy; Clinical Response; Pathological Response
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simvastatin (Experimental): The group received standard treatment with simvastatin 40mg in capsule by oral route, once a day, for 21 days (every cycle of the chemotherapy regiment)
  Interventions: Drug: Simvastatin 40mg
- Placebo (Placebo Comparator): The group received standard treatment with placebo 40mg in capsule by oral route, once a day, for 21 days (every cycle of the chemotherapy regiment)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Simvastatin 40mg — The administration of Simvastatin 40 mg in addition to ACT regiment of neoadjuvant chemotherapy
  Other Names: Simvastatin
  Arms: Simvastatin
Drug: Placebo — The administration of Placebo capsule 40 mg in addition to ACT regiment of neoadjuvant chemotherapy
  Other Names: Placebo oral capsule 40 mg
  Arms: Placebo

SUMMARY:
Introduction: Most cases of Triple Negative Breast Cancer (TNBC) have a high proliferation rate. TNBC is associated with a poor prognosis, a high recurrence rate, and a high incidence of distant metastases. The Epithelial-Mesenchymal Transition process (EMT) plays an essential role in the metastatic process. EMT markers were also more abundant in TNBC and contributed to a poorer TNBC prognosis. As an important EMT marker, the increased expression of vimentin also contributed to the increase in TNBC aggressiveness and resistance to chemotherapeutic agents. Through the mechanism of action in inhibiting the mevalonate pathway, statins can help inhibit the EMT process in metastases. Notably, simvastatin promotes the down-regulation of vimentin in breast cancer cells. The combination of statins and neoadjuvant chemotherapy (NAC) improves the cancer patient's response. This study is expected to evaluate the role of a combination between NAC and simvastatin on therapeutic response in TNBC patients through vimentin expression.

Methods: This study is a double-blind, randomized, placebo-controlled trial conducted in Dr. Cipto Mangunkusumo National Central General Hospital. An expected total of 26 TNBC patients will be assessed for eligibility and asked for informed consent. Patients with the plan to have ACT (Doxorubicin hydrochloride, Cyclophosphamide, Paclitaxel) chemotherapy regimen will receive either a combination of ACT-Simvastatin (40 mg/day) or ACT-Placebo. The biopsy will be taken pre-NAC to make the histopathological diagnosis and examine the expression of vimentin. Patients will be evaluated for adverse effects reaction every cycle and the clinical response after 8 cycles. The post-intervention biopsy will be conducted after the cycle finish. The pathological response and vimentin expression will be reviewed from the obtained samples.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients with advanced breast cancer (locally advanced and distantly advanced) with triple-negative molecular type confirmed by biopsy and immunohistochemical examination.
2. The patient planned to receive 8 cycles of AC-T chemotherapy.
3. Patient age > 18 years.
4. Willing to participate in research by signing informed consent.

Exclusion Criteria:

1. The patient is pregnant or breastfeeding.
2. Patients who have received chemotherapy or are on simvastatin therapy.
3. Allergy to statins.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-08-19 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Vimentin Expression | 6 months
  Vimentin expression is measured based on Histoscore (H-Score) with immunohistochemistry examination:
  * 0-50 : negative (0)
  * 51-100 : weak positive (1+)
  * 101-200 : moderate positive (2+)
  * 201-300 : strong positive (3+)

SECONDARY OUTCOMES:
Pathological Response | 6 months
  Pathological Response as Measured by Miller-Payne system
  Evaluation before and after chemotherapy, divided into:
  1. Grade 1: There is no significant change or reduction in cancer cells.
  2. Grade 2: Reduction of <30% cancer cells
  3. Grade 3: Reduction of cancer cells between 30-90%
  4. Grade 4: Reduction of > 90% cancer cells
  5. Grade 5 : There are no residual cancer cells. DCIS (Ductal Carcinoma In Situ) might be detected.
Clinical Response | 6 months
  Clinical response based on WHO (World Health Organization) criteria:
  1. Complete Response (CR): Disappearance
  2. Partial Response (PR): 50% decrease
  3. Stable Disease(SD): Neither PR nor PD criteria met
  4. Progressive Disease (PD):25% increase; no CR, PR, or SD documented before increased disease

CONTACTS AND LOCATIONS:
Overall Officials: Erwin D Yulian, MD, Principal Investigator — Surgical Oncology Division, Department of Surgery, Universitas Indonesia; Tantri Hellyanti, MD, Study Director — Department of Pathological Anatomy, Universitas Indonesia; Shabrina Adzania, MD, Study Chair — Research Assistant, Department of Surgery, Universitas Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo National Central General Hospital, Jakarta Pusat, DKI Jakarta, Indonesia